CLINICAL TRIAL: NCT05899621
Title: A Real-world Study of the Efficacy and Safety of Obinutuzumab-based Therapy for Previously Untreated Follicular Lymphoma
Brief Title: A Real-world Study of Obinutuzumab-based Therapy for Previously Untreated FL
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department Affiliation: Ruijin Hospital, Ruijin Hospital
Other Study IDs: FL-Gbased
Record Dates: First submitted 2023-05-01; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Follicular Lymphoma
Keywords: obinutuzumab; Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — obinutuzumab; Lenalidomide; Bendamustine Hydrochloride; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GR: Induction(six 21-day cycles): obinutuzumab (G), 1000mg, IV, D1/8/15 (C1), D1 (C2-6); lenalidomide (R), 25mg, PO, D2-11; Maintenance: obinutuzumab (G), 1000mg, every 3 months for 2 years; lenalidomide (R), 25mg, PO, D1-10, every 28 days for 6 cycles
  Interventions: Drug: Obinutuzumab; Drug: Lenalidomide
- GB: Induction(six 21-day cycles): obinutuzumab (G) 1000mg, IV, D1/8/15 (C1), D1 (C2-6); bendamustine (B), 90 mg/m2, IV, D1-2; Maintenance: obinutuzumab (G), 1000mg, IV, every 3 months for 2 years
  Interventions: Drug: Obinutuzumab; Drug: Bendamustine
- GCHOP: Induction(six 21-day cycles): obinutuzumab (G), 1000mg, IV, D1/8/15 (C1), D1 (C2-6); prednisone (P), 100 mg, PO, D1-5；cyclophosphamide (C), 750 mg/m2, IV, D1; vincristine (O), 1.4 mg/m2 (maximum 2 mg), IV, D1; doxorubicin (H), 50 mg/m2, IV, D1; Maintenance: obinutuzumab (G), 1000mg, IV, every 3 months for 2 years
  Interventions: Drug: Obinutuzumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Lenalidomide — Lenalidomide PO will be administered as per the schedule specified in the respective arm.
  Groups: GR
Drug: Bendamustine — Bendamustine IV infusion will be administered as per the schedule specified in the respective arm.
  Groups: GB
Drug: Cyclophosphamide — Cyclophosphamide IV infusion will be administered as per the schedule specified in the respective arm.
  Groups: GCHOP
Drug: Doxorubicin — Doxorubicin IV infusion will be administered as per the schedule specified in the respective arm.
  Groups: GCHOP
Drug: Vincristine — Vincristine IV infusion will be administered as per the schedule specified in the respective arm.
  Groups: GCHOP
Drug: Prednisone — Prednisone PO will be administered as per the schedule specified in the respective arm.
  Groups: GCHOP

SUMMARY:
This study aims to observe and explore the efficacy and safety of obinutuzumab-based therapy for previously untreated follicular lymphoma

DETAILED DESCRIPTION:
This study aims to observe and explore the efficacy and safety of obinutuzumab-based therapy for previously untreated follicular lymphoma. This study is a non-interventional real world, observational study and all registered data are collected from real clinical practice cases. The medical data includes patient demographic, tumor characteristics, laboratory examination, history of treatments, adverse reactions, efficacy results and possible prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed CD20 positive follicular lymphoma grade 1, 2, or 3A based on 2016 WHO classification
* Treatment naive
* Age ≥ 18 years
* Indications for treatment confirmed
* Must has measurable lesion in CT or PET-CT prior to treatment
* Considered suitable for GR, GB or GCHOP regimens
* Informed consented

Exclusion Criteria:

* Transformed follicular lymphoma or 3B follicular lymphoma;
* HBsAg positive and / or HBcAb positive with HBV DNA titer; HCV antibody positive with HCV-RNA; or HIV positive
* Central nervous system or meninges involved
* Any drug contraindication in the treatment plan
* Patients judged by other researchers to be unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients age ≥18 years with grade 1 to 3a FL.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | End of treatment visit (6 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Complete response rate (CR) | End of treatment visit (6 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of first treatment until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Duration of response | Baseline up to data cut-off (up to approximately 2 years)
  Time from first occurrence of documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR. Tumor assessments were performed with PET-CT.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No